CLINICAL TRIAL: NCT07206563
Title: Penfluridol for Relapsed/Refractory Small Cell Lung Carcinoma and Small Cell Cervical Cancer: An Open-Label, Multicenter, Single-Arm Ib/II Trial
Brief Title: Penfluridol for Relapsed/Refractory Small Cell Cancers
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT250646
Record Dates: First submitted 2025-09-16; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Small Cell Carcinoma; Small Cell Carcinoma of Lung; Small Cell Lung Cancer ( SCLC ); Small Cell Cervical Carcinoma
Keywords: Small cell cervical carcinoma; small cell lung carcinoma; Relapsed/refractory; Phase Ib/II; DRD2 targeting
MeSH Terms: conditions — Carcinoma, Small Cell; Small Cell Lung Carcinoma; Recurrence | interventions — Penfluridol

STUDY DESIGN:
Intervention Model Description: Ultra-rare population
  * Cervical small-cell carcinoma accounts for <2 % of all cervical cancers, and third-/later-line SCLC represents <5 % of lung-cancer cases.
  * A randomized study would require prohibitively large sample sizes and prolong accrual beyond the 3-year funding window.
  Absence of an established active comparator
  * Historical controls (retrospective cohorts) show ORR ≤ 12-18 % and median PFS ≤ 2.5 months in ≥3-line therapy.
  * No standard-of-care regimen is approved after ≥2 prior systemic treatments, making a placebo or active-control arm ethically questionable.
  Signal-seeking objective
  * The primary goal of this first-in-class oncology application is to define the recommended Phase II dose (RP2D) and to estimate preliminary efficacy signals (ORR), not to demonstrate superiority.
  * A single-arm design with an explicit Simon two-stage rule (H0: ORR ≤ 10 % vs. H1: ≥15 %) provides the most efficient path to accept or reject further development with ≤33 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penfluridol Monotherapy for Relapsed/Refractory Small-Cell Lung or Cervical Cancer (Experimental): Intervention: Penfluridol, an oral antipsychotic drug, is used as monotherapy. It targets DRD2, inhibits glycolysis, and induces apoptosis.
  Dosing Schedule:
  Phase Ib: 3+3 dose-escalation design. Initial dose 20 mg weekly, escalating to 40 mg, then 60 mg until recommended Phase II dose (RP2D) is determined based on 21-day DLT assessment.
  Phase II: Expansion cohort at RP2D to further evaluate safety and estimate ORR. Duration: Treatment continues until progression, unacceptable toxicity, withdrawal, or investigator decision.
  Monitoring: Regular AE/SAE monitoring using NCI-CTCAE v5.0. Assessments include weekly vital signs, biweekly blood tests, and ECGs every 2 weeks. Tumor response evaluated by RECIST 1.1 criteria with imaging every 2-3 cycles.
  Dose Modification: Adjustments made for EPS, QTc prolongation, and proteinuria. Rationale for Single-Arm Design: Chosen due to the ultra-rare patient population and lack of established comparators. Efficient for determining RP2D and ORR.
  Interventions: Drug: Penfluridol Monotherapy for Relapsed/Refractory Small-Cell Lung or Cervical Cancer

INTERVENTIONS:
Drug: Penfluridol Monotherapy for Relapsed/Refractory Small-Cell Lung or Cervical Cancer — Intervention: Penfluridol, an oral antipsychotic drug, is used as monotherapy. It targets DRD2, inhibits glycolysis, and induces apoptosis.
  Dosing Schedule:
  Phase Ib: 3+3 dose-escalation design. Initial dose 20 mg weekly, escalating to 40 mg, then 60 mg until recommended Phase II dose (RP2D) is determined based on 21-day DLT assessment.
  Phase II: Expansion cohort at RP2D to further evaluate safety and estimate ORR. Duration: Treatment continues until progression, unacceptable toxicity, withdrawal, or investigator decision.
  Monitoring: Regular AE/SAE monitoring using NCI-CTCAE v5.0. Assessments include weekly vital signs, biweekly blood tests, and ECGs every 2 weeks. Tumor response evaluated by RECIST 1.1 criteria with imaging every 2-3 cycles.
  Dose Modification: Adjustments made for EPS, QTc prolongation, and proteinuria. Rationale for Single-Arm Design: Chosen due to the ultra-rare patient population and lack of established comparators. Efficient for determining RP2D and ORR.
  Other Names: Semap; R-16341

SUMMARY:
Penfluridol for Relapsed/Refractory Small-Cell Carcinoma of the Lung or Cervix: A Multicenter, Open-Label, Single-Arm Phase Ib/II Trial This study evaluates the safety and anti-tumor activity of oral penfluridol, a first-generation antipsychotic that pre-clinically inhibits small-cell carcinoma (SCC) growth via DRD2 blockade, metabolic reprogramming and apoptosis induction. After ≥2 prior systemic regimens, 33 adult patients (18-75 y) with measurable, metastatic or recurrent lung or cervical SCC will be enrolled across five Chinese centers. A 3+3 dose-escalation (Ib) will establish the recommended Phase II dose (RP2D); an expansion cohort (II) will examine objective response rate (ORR, RECIST 1.1). Secondary end-points include duration of response, progression-free survival, overall survival, safety and exploratory biomarkers. Key inclusion: ECOG 0-1, adequate organ function, no active brain metastases. Penfluridol is administered once weekly, dose-escalated from 20 mg to RP2D, continued until progression or intolerance. Patients receive free study drug, PET imaging and laboratory monitoring.

DETAILED DESCRIPTION:
Rationale and Preclinical Justification Small-cell carcinoma of the lung (SCLC) and cervix (SCCC) represent aggressive malignancies with a paucity of effective therapeutic options upon relapse, leading to dismal survival outcomes. To address this unmet need, a high-throughput drug screening was conducted utilizing patient-derived organoid (PDO) models of SCLC and SCCC. This screening identified penfluridol, a first-generation antipsychotic drug with a long-established human safety profile, as a potent inhibitor of small-cell carcinoma growth. Its anti-tumor efficacy is mechanistically attributed to dual pathways: 1) antagonism of dopamine receptor D2 (DRD2), a target implicated in cancer stem cell maintenance and proliferation, and 2) induction of metabolic stress via inhibition of glycolysis, leading to AMPK/FOXO3a-mediated apoptosis. Notably, penfluridol's inherent ability to penetrate the blood-brain-barrier positions it as a potential therapeutic candidate for addressing the common site of metastasis in SCLC. This study aims to clinically reposition penfluridol based on this compelling preclinical evidence.

Study Design and Technical Considerations This is an open-label, multicenter, seamless Phase Ib/II trial. The design integrates a dose-finding phase followed by an efficacy expansion phase to efficiently evaluate both safety and preliminary activity.

Phase Ib (Dose Escalation): Utilizes a standard 3+3 design to determine the Recommended Phase II Dose (RP2D). The starting dose is 20 mg orally once weekly, with planned escalation to 40 mg and 60 mg. The RP2D will be defined as the highest dose at which ≤1 of 6 patients experiences a dose-limiting toxicity (DLT) during the first 21-day cycle. Pharmacokinetic profiling will be performed to characterize exposure at each dose level.

Phase II (Expansion Cohort): Aims to estimate the objective response rate (ORR) at the RP2D. The study employs a Simon's two-stage minimax design to test the null hypothesis that the true ORR is ≤10% against an alternative of ≥30%, with 90% power and a one-sided alpha of 0.05. This design allows for early termination for futility.

Biomarker Strategy: The protocol incorporates a comprehensive exploratory biomarker plan. This includes correlative analyses of DRD2 expression in archival tumor tissue, serial monitoring of cell-free DNA (cfDNA) for dynamic changes in tumor burden, and assessment of metabolic response via FDG-PET imaging to elucidate potential biomarkers of response and resistance.

Safety Monitoring Focus Given penfluridol's known safety profile from psychiatric use, the protocol institutes enhanced, protocol-specified monitoring for specific risks. This includes regular assessments for extrapyramidal symptoms (using the RSESE scale) and rigorous cardiac monitoring (serial ECGs for QTc interval assessment) beyond standard CTCAE reporting. An independent Data Monitoring Committee (IDMC) will review accumulating safety and efficacy data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 75 years, inclusive, regardless of gender.
2. Histologically or cytologically confirmed small-cell carcinoma of the lung or cervix that is not curable by surgery or radiochemotherapy.
3. Have received at least two prior systemic treatment regimens, including etoposide and platinum-based chemotherapy, and have experienced disease progression.
4. No receipt of investigational or approved cytotoxic chemotherapy within 28 days before enrollment; no receipt of alkylating agents within 42 days before enrollment; no receipt of investigational or approved targeted therapy within 28 days or 5 half-lives before enrollment (whichever is shorter, but not less than 14 days); no radiotherapy within 14 days before enrollment.
5. Presence of measurable disease according to RECIST 1.1 criteria; measurable lesions are defined as lesions that can be accurately measured in at least one dimension (longest diameter ≥10 mm on CT or MRI scans, and lymph nodes with short-axis diameter ≥15 mm).
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Expected survival of ≥12 weeks.
8. Recovery of prior anticancer treatment toxicities to ≤Grade 1 (except for alopecia, pigmentation, or other toxicities deemed non-safety risks by the investigator); for irreversible toxicities that are not expected to worsen with study drug administration (e.g., hearing loss), inclusion may be considered after consultation with the medical monitor. Recovery of peripheral neuropathy to ≤Grade 2 after prior use of cisplatin or etoposide may be considered for inclusion after consultation with the medical monitor. For late toxicities caused by radiotherapy that cannot be recovered, inclusion may be considered after consultation with the medical monitor.
9. Laboratory tests: Absolute neutrophil count ≥1.5×10⁹/L; platelets ≥75×10⁹/L; hemoglobin ≥90 g/L; serum creatinine ≤1.5 times the upper limit of normal (ULN); urine protein <2+ or 24-hour urine protein <1.0 g; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times ULN (or ≤5 times ULN in the presence of liver metastasis); total bilirubin ≤1.5 times ULN; albumin ≥28 g/L; coagulation function: prothrombin time (PT) and international normalized ratio (INR) ≤1.5×ULN.
10. Female subjects with negative urine or blood HCG (except for menopausal and hysterectomy cases); sexually active female subjects and their partners must agree to use effective contraception (e.g., combined hormonal contraception, intrauterine device, bilateral tubal ligation, vasectomy, abstinence) during the study and for 6 months after the last dose.
11. Availability of tumor specimens (paraffin-embedded blocks or frozen tissue) from prior resection or biopsy sufficient for pharmacodynamic assays (≥3 slides for immunohistochemistry IHC) (mandatory for dose-expansion cohort patients only).
12. Ability to understand the study and voluntary consent to participate in the trial by the patient or their legal representative, with signed informed consent.

Exclusion Criteria:

1. Histological diagnosis of squamous cell carcinoma, adenocarcinoma, or other non-small-cell types of lung or cervical cancer.
2. Concurrent enrollment in another clinical trial, unless it is an observational, non-interventional study or the follow-up period of an interventional study.
3. Known hypersensitivity to any component of penfluridol or similar compounds with comparable chemical or biological properties.
4. Prior exposure to penfluridol.
5. Known presence of leptomeningeal metastasis, spinal cord compression, leptomeningeal disease, or active brain metastases. However, patients with asymptomatic brain metastases (no neurological deficits, seizures, or other typical symptoms and signs of central nervous system metastasis; no requirement for corticosteroids) or those who have been treated and are stable on imaging for at least 4 weeks before study treatment (with no new or enlarged brain metastases) and have discontinued systemic corticosteroids and anticonvulsant medications for at least 2 weeks may be included.
6. Uncontrolled comorbid conditions, including but not limited to persistent or active infections or psychiatric/social conditions that would limit compliance with study requirements.
7. Positive for human immunodeficiency virus (HIV) on combination antiretroviral therapy.
8. Cardiovascular history or comorbidities: Known history of arrhythmias (including atrial fibrillation, tachycardia, or bradycardia), except for benign ventricular premature beats; history of CHF, MI, or stroke within the past 3 months.
9. History of seizure within the past 3 months.
10. Gastrointestinal dysfunction or disease that may significantly alter the absorption of penfluridol (e.g., uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
11. Known history of allogeneic organ transplant or allogeneic hematopoietic stem cell transplant.
12. Uncontrolled severe medical conditions that, in the opinion of the investigator, would affect the patient's ability to receive the study treatment, such as severe internal medicine conditions, including hepatic or renal insufficiency, severe cardiovascular disease, cerebrovascular disease, uncontrolled diabetes, or uncontrolled infections.
13. Pregnant or breastfeeding women; sexually active female subjects unwilling to use contraception.
14. Presence of symptomatic or unstable pleural effusion, ascites, or pericardial effusion requiring repeated drainage.
15. Patients deemed unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dose (RP2D) of penfluridol [Phase Ib] | From the first dose until the completion of the DLT observation period (21 days) for the first cohort of patients at each dose level (The Phase Ib dose-escalation stage is anticipated to take approximately 9 months).
  To determine the Recommended Phase II Dose (RP2D) of oral penfluridol for the treatment of relapsed/refractory small cell lung cancer and small cell cervical cancer.
Objective Response Rate (ORR) [Phase II] | From the first dose of study drug until disease progression, start of new anticancer therapy, or death from any cause (whichever occurs first), assessed up to approximately 24 months.
  To evaluate the antitumor activity of oral penfluridol at the RP2D as measured by the Objective Response Rate.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From the first dose of study drug until 30 days after the last dose, assessed up to approximately 24 months.
  To evaluate the safety and tolerability profile of oral penfluridol.
Duration of Response (DOR) | From the first documented objective response until disease progression or death (whichever occurs first), assessed up to approximately 24 months.
  To assess the durability of tumor responses.
Progression-Free Survival (PFS) | From the first dose until disease progression or death (whichever occurs first), assessed up to approximately 24 months.
  To assess disease control.
Overall Survival (OS) | From the first dose until death from any cause, assessed up to approximately 36 months.
  To evaluate the overall survival benefit.
Disease Control Rate (DCR) | From the first dose until documented disease progression, assessed up to approximately 24 months.
  To evaluate the proportion of patients achieving disease control.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Wu, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No